CLINICAL TRIAL: NCT02283281
Title: Effects of a Cannabis Extract as Anaesthetic Premedication on Postoperative Pain, Nausea-vomiting and Perioperative Anxiety
Brief Title: Anesthetic Premedication With a Cannabis Extract (Cannapremed)
Acronym: Cannapremed
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cannapremed-HMO-CTIL
Record Dates: First submitted 2014-11-02; First posted 2014-11-05 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting; Anxiety
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Anxiety Disorders | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cannabis oil high dose (Experimental): Single-dose, before anesthetic induction: 21.6 mg tetrahydrocannabinol + 20 mg cannabidiol, Sub-linguistic
  Interventions: Drug: Tetrahydrocannabinol
- Cannabis oil low dose (Experimental): Single-dose, before anesthetic induction: 10.8 mg tetrahydrocannabinol + 10 mg cannabidiol, Sub-linguistic.
  Interventions: Drug: Tetrahydrocannabinol
- Control (Placebo Comparator): Single-dose, before anesthetic induction: Dummy oromucosal spray containing alcohol vehicle without Cannabis oil .
  Interventions: Drug: Dummy oromucosal

INTERVENTIONS:
Drug: Tetrahydrocannabinol — 1:1 THC to CBD standardized extract from cannabis plant
  Other Names: Cannabis oil
  Arms: Cannabis oil high dose; Cannabis oil low dose
Drug: Dummy oromucosal — drops containing only Olive oil vehicle without the active compound (i.e.: without Cannabis oil)
  Other Names: Cannabis oil placebo
  Arms: Control

SUMMARY:
Clinical evidence about the effects of cannabis in a perioperative setting or for the management of acute pain is rather scarce, mostly consisting of case report-based opinions on adverse events during or after general anesthesia after smoking cannabis, experimental pain trials in healthy volunteers, and a few clinical trials using different drugs, dosages and routes of administration. It is difficult to draw strong conclusions from the available evidence, that may seem sometimes even contradictory, mainly due -the investigators believe- to the many sources of variability in the study designs (e.g.: heterogeneity of the study samples, underpowered, unblinding, lack of randomization, timing of the therapeutic intervention, different experimental pain models, inclusion of different kind of surgical pain, etc.). Nevertheless, expert's opinion after a critical review of the literature is that cannabis and cannabinoids may have a beneficial role in the management of acute post-operative pain and nausea, at least for a selected group of patients and through an appropriate therapeutic intervention.

Therefore, it seems to us pertinent to carry out an investigation in order to re-evaluate the issue of perioperative cannabis use through a sufficiently powered and controlled clinical trial. Some of cannabis effects such as sedation, bronchodilation, dryness of respiratory secretions, vein dilation, and increase of heart rater without producing hypertension, make of it an attractive option for pre-medication; while its antiemetic properties and its analgesic potential without causing respiratory depression may be profitable for the post-operative period.

Cannabis oil seem to be most suitable to our investigation. The co-administration of tetrahydrocannabinol (THC) with cannabidiol (CBD) may translate into additional therapeutic benefits with an attenuation of adverse effects. The investigators expect to obtain less sedation, milder "high", lower incidence of anxiety, tachycardia, and hyperalgesia, as compared with THC-only acute pain trials.

DETAILED DESCRIPTION:
The selection of patients will be done during the pre-anesthetic assessment the day before surgery. After obtaining informed consent, eligible patients will be randomly allocated to one of the following regimes: Cannabis oil high dose (21.6 mg THC + 20 mg CBD), Cannabis oil low dose (10.8 mg THC + 10 mg CBD), placebo control (no premedication drugs).

Treatments will be administered in a double-dummy manner. Identical bottles of Cannabis oil and placebo should be obtained from the manufacturer (Bazelet group). Identical prefilled vials containing sodium Olive oil should be prepared by the hospital pharmacist. To the best of our knowledge, no clinical studies evaluating the effects of Cannabis oil on acute pain or in a perioperative setting have been done to date. Therefore, the investigators estimate a Cannabis oil dose range that seems reasonable to obtain relevant clinical and a manageable occurrence of adverse events, mainly based on the recommendations from the manufacturer, on the available pharmacological data presented in the previous section and on the results of other clinical trials with a similar design using comparable doses of oral THC. Nevertheless, the first 10 patients will be randomly assigned either to the Cannabis oil low dose group or to the placebo control group only. The investigators will proceed with the full four-group randomization only if no serious adverse events are registered among the 10 first recruited patients.

At the arrival to the operating room, blood samples for baseline levels of cannabinoids will be drawn at the moment of placing the intravenous line, and the first anxiety assessment should be done by the examiner/anesthetist. The study drugs will be administered at the entrance to the O.R. or at the induction room 15 minutes before the induction of anesthesia (i.e.:). Premedication dose should be calculated to be the equivalent of 10 mg and 20 mg oral THC for the low and high dose groups, respectively (4, 8 puffs). At the same time, the prefilled drops containing Olive oil will be administered as intravenous bolus. The patients will be immediately connected to the standard O.R. monitoring.

Induction of general anaesthesia will be done in a standardized fashion with fentanyl 2 µg/Kg, propofol 1-4 mg/Kg (and vecuronium 0.1 mg/Kg if intubation is required). For anaesthetic maintenance, isoflurane 0.7-2% on 1:2 oxygen : nitrous oxide gas mixture, and fentanyl boluses 1 µg/Kg to keep a bispectral index (BIS) between 40 to 60, and a heart rate and mean arterial pressure between 70-130% from pre-induction baselines. Preemptive antiemetics (e.g.: granisetron, ondansetron, metoclopramide, dexamethasone, etc.) should not be given. No additional analgesics should be administered (e.g.: ketorolac or other NSAID's, dipyrone).

A loading dose of morphine 0.2 mg/Kg will be given before the end of surgery provided that the patient can maintain spontaneous breathing or pressure support ventilation. Intravenous morphine patient-controlled analgesia (PCA) will be initiated on the arrival to the recovery room with boluses of 1 mg and a lockout time of 6 minutes, without background.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgeries suitable for postoperative pain treatment with intravenous morphine patient-controlled analgesia.
* American Society of Anesthesiologist (ASA) risk I or II

Exclusion Criteria:

* ASA III or higher
* Cannabis use within the last 6 months
* Pregnancy
* Emergency surgeries
* Regional anesthesia
* Ischemic heart disease
* Renal failure
* History of psychosis
* Cognitive impairment or inability to answer questions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain - VAS | 24 hours
  Self-reported visual analog scale (VAS 0 - 100 mm) at rest and on movement. Pre-operative baseline, on arrival to recovery room, after 1 h, before discharge, at 6, 12, and 24 h.
Postoperative pain - PCA | 24 hours
  Count of patient-controlled analgesia pushes 1 hour after arrival to the recovery room, before discharge, at 6, and 12.
  Total dose of morphine received in 24 hours.

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) score | 24 hours
  PONV score (0 - 4) on arrival to recovery room, after 1 hour, before discharge, at 6, 12, and 24 hours.
  0. No nausea
  1. Nausea sometimes
  2. Nausea most of the time
  3. Dry retching or vomiting
  4. Dry retching or vomiting twice or more
Anxiety - VAS | 6 hours
  Self-assessed anxiety visual analog scale (0-100 mm) on arrival to the OR; on arrival to and before discharge from recovery room.
Cannabinoid blood levels | 24 hours
  Blood sampling from arterial line inserted on arrival to the OR before the main premedication dose, after 30 min, at 1, 3, 6, 12, and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Elyad Davidson, M.D., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hasassah - Hebrew University Ein Kerem Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laursen DR, Nejstgaard CH, Bjorkedal E, Frost AD, Hansen MR, Paludan-Muller AS, Prosenz J, Werner CP, Hrobjartsson A. Impact of active placebo controls on estimated drug effects in randomised trials: a systematic review of trials with both active placebo and standard placebo. Cochrane Database Syst Rev. 2023 Mar 6;3(3):MR000055. doi: 10.1002/14651858.MR000055.pub2. PMID 36877132